CLINICAL TRIAL: NCT04537819
Title: A Multicenter, Randomized, Open, Comparative Study of Efficacy, Safety and Tolerability of Imupret Application in the Concept of Delayed Prescription of Antibiotics in Children, Aged 6-12 With Acute Tonsillitis
Brief Title: Study of Imupret Application in the Technology of Delayed Prescription of Antibiotics in Patients With Acute Tonsillitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivano-Frankivsk National Medical University (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATi-2
Record Dates: First submitted 2020-07-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Acute Tonsillitis
Keywords: Acute tonsillitis; antibiotics; phytotherapy
MeSH Terms: interventions — imupret

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The main group (Experimental): 1. soft diet; 2. Elimination of factors that irritate the mucous membrane of the pharynx (thermal, chemical); 4. Local NSAIDs - benzydamine hydrochloride. 5. Imupret oral drops in the age-related dosage of 6 times per day for 6 days with the subsequent transition to the regime of 15 drops / 3 times in a day according to the patient's condition.
  6. Paracetamol as antipyretic, if necessary.
  Interventions: Drug: Imupret in addition to local NAID
- The comparison group (Other): 1. soft diet; 2. Elimination of factors that irritate the mucous membrane of the pharynx (thermal, chemical); 4. Local NSAIDs - benzydamine hydrochloride. 5. Paracetamol as antipyretic, if necessary.
  Interventions: Drug: Local NAID (Benzydamin)

INTERVENTIONS:
Drug: Imupret in addition to local NAID — Additional prescription of Imupret oral drops to conventional therapy with local NAID (Benzydamine hydrochloridy), elimination of irritating factors in the diet and acetaminophen (if necessary)
  Other Names: BNO 1030 extract from 7 plants (active substance of Imupret)
  Arms: The main group
Drug: Local NAID (Benzydamin) — (Benzydamine hydrochloridy) and acetaminophen (if necessary), elimination of irritating factors in the diet
  Other Names: Tantum Verde
  Arms: The comparison group

SUMMARY:
The problem of acute tonsillitis (AT) is one of the most urgent in modern clinical medicine. The prevalence of pathology ranges from 2 to 15% of the total population.

AT (ICD J03.0-J03.9) in most cases is due to viral infections. Bacterial acute tonsillitis occurs in immunocompetent children in 20-30% of cases.

To determine the indications for antibacterial therapy, the Mclsaac scale is a commonly used tool for decision. This scale is used to classify patients according to their symptoms and to determine the patients for whom antibiotic therapy is not indicated.

Thus, in most cases of acute tonsillitis (even if there are 4-5 points according to the scale), it has to be taken into account that there is a low probability of the presence of GABS. Therefore, there are no unconditional indications for the prescription of antibiotics. Unjustified antibiotic therapy of AT plays a significant role in the formation of antibiotic resistance.

To prevent unjustified prescription of antibiotics, a therapeutic concept of delayed administration is proposed. A patient with AT is prescribed treatment with antibiotics in a delayed manner. In the absence of a positive effect within 36-48 hours from the beginning of treatment with Imupret, the antibacterial therapy is started. The advantage of deferred antibiotic prescription is, that a higher number of patients and doctors, awaiting antibiotic therapy, may be more agreeable with this way of treatment than with a complete rejection of the antibiotic's prescription. So delayed use of antibiotics is an important treatment strategy to reduce the number of unreasonable prescriptions of antibiotics.

Considering this fact, it becomes necessary to use drugs with a complex effect and evidence-based efficacy base for acute tonsillitis. At the moment, there is an insignificant evidence base for the application of the phytoneering drug Imupret in acute tonsillitis. The spectrum of its pharmacological properties includes antiviral, antibacterial, anti-inflammatory, and immunomodulating effects. The combination of these properties makes it possible to influence practically all parts of acute tonsillitis. The already existing studies were not conducted under GCP conditions. Confirmation of the high effectiveness of Imupret in the treatment of acute tonsillitis would serve as a rationale for optimizing the treatment regimen of this nosology and recommendations for the inclusion of the drug in national guidelines.

DETAILED DESCRIPTION:
Study of Therapeutic Efficacy, Safety, and Tolerability of Imupret application in the therapeutic concept of delayed prescription of antibiotics in patients with severe acute tonsillitis in children, aged 6-12.

Acute tonsillitis in most cases is due to viral infections. Bacterial tonsillitis occurs in immunocompetent children in 20-30% of cases, adults - in 5-15%, and the most frequent cause of it is β-hemolytic streptococcus group A (GABS).

Acute tonsillitis is defined as the sudden appearance of the following symptoms: sore throat, hyperemia, edema of the tonsils, increase in swollen lymph nodes, and non-specific additional symptoms like fever, weakness, and joint pain. There are no pathognomonic symptoms of bacterial tonsillitis. To assess the patient's condition and to determine the indications for antibacterial therapy, the Mclsaac scale is a commonly used tool for decision. This scale is used to classify patients according to their symptoms and to determine the patients for whom antibiotic therapy is not indicated.

McIsaac scale (sum of scores) The probability of the identification of β-hemolytic streptococcus in a smear from pharynx -1 or 0 - 1% 1-10% 2 ~17% 3 ~35% 4 or 5 ~50% Thus, in most cases of acute tonsillitis (even if there are 4-5 points according to the scale), it must be considered that there is a low probability of the presence of GABS. Therefore, there are no unconditional indications for the prescription of antibiotics.

Unjustified antibiotic therapy of acute tonsillitis based on "sore throat" or "exudate (plaque) tonsils" only does not affect pain and lads the formation of antibiotic resistance. In order to avoid the irrational use of antibiotics, one should distinguish the desire of the patient or his parents to get rid of the pain, from the rational assessment of the doctor for all pros and cons about an antibacterial therapy.

To prevent the unjustified prescription of antibiotics, a therapeutic concept of delayed administration is proposed. A patient with acute tonsillitis is prescribed treatment with antibiotics in a delayed manner. In the absence of positive dynamics within 36-48 hours from the beginning of treatment with Imupret the antibacterial therapy is started. The advantage of deferred antibiotic prescription is, that a higher number of patients and doctors, awaiting antibiotic therapy, may be more agreeable with this way of treatment than with a complete rejection of the antibiotic's prescription. Therefore, the delayed use of antibiotics is an important treatment strategy to reduce the number of unreasonable prescriptions of antibiotics.

Considering this fact, it becomes necessary to use drugs with a complex effect on the main processes of pathogenesis and have an evidence-based efficacy for acute tonsillitis. Now, there is an insignificant evidence base for the application of the herbal drug Imupret in acute tonsillitis. The spectrum of its pharmacological properties includes antiviral, antibacterial, anti-inflammatory, and immunomodulating effects. Additionally, a good safety profile allows to consider Imupret as an adequate basic therapy for the treatment of acute tonsillitis in the therapeutic concept of delayed prescription of antibiotics. The already existing studies were not conducted under GCP conditions. Confirmation of the high effectiveness of Imupret in the treatment of acute tonsillitis would serve as a rationale for optimizing the treatment regimen of this nosology.

Proposed trial design: open-label, exploratory, comparative, multicenter, randomized, prospective, parallel-group study.

Treatment:

The comparison group (n = 100): soft diet; elimination of factors that irritate the mucous membrane of the pharynx (thermal, chemical); local NSAIDs - benzydamine hydrochloride (Tantum Verde); acetaminophen as antipyretic if necessary.

The main group (n=100): soft diet; elimination of factors that irritate the mucous membrane of the pharynx (thermal, chemical); local NSAIDs - benzydamine hydrochloride; Imupret oral drops in the age-related dosage of 6 times per day for 6 days with the subsequent transition to the regime of 15 drops / 3 times in a day according to the patient's condition; acetaminophen as antipyretic, if necessary.

Schedule of visits. During the study, 3 planned visits: Visit 1 (The 1-st day): screening, randomization, and treatment; evaluation by Mc Isaac Score scale; LTM Scale (Local Tonsillitis Manifestation Scale): (5 symptoms: Sore throat at swallowing (0 - absent, 1 - mild, 2 - moderate, 3 - severe / pronounced); Sore throat at rest; Throat irritation at rest; Palatine tonsils hyperemia; Palatine tonsils edema); Patients self-assessment (VAS; 0-10). Visit 2 (3rd±1 day): intermediate evaluation of the effectiveness of treatment - clarification of the patient's condition, the need to prescribe an antibiotic; evaluation by LTM Scale, patients' self-assessment (VAS; 0-10). Visit 3: intermediate evaluation of the effectiveness of treatment (day 5-day ±1) via telephone (or visit if necessary); patients' self-assessment (VAS; 0-10). Visit 4: final (10th day ±1 day). Evaluation by LTM Scale (0-15), patients' self-assessment (VAS; 0-10). 5 Follow up; day 28: evaluation of the long-term effects of treatment.

An unscheduled visit can be made if the patient's condition worsens (according to the patient and/or the researcher, including if the symptoms of the disease persist or worsen, including but not limited to an increase in the temperature in the armpit above 38.0 ° C at the 3rd and/or subsequent days of treatment).

The total duration of the treatment: 10 days. The total duration of the study for one patient is no longer than 38 days.

Objectives of the study: To investigate the influence of Imupret prescriptions in the therapeutic concept of delayed prescription of antibiotics to:

* need for antibiotics;
* regression of the tonsillitis symptoms;
* duration of antipyretics administration.

Proposed parameters of interest:

* The severity of symptoms of tonsillitis, on the Visit 2 compared to the Visit 1. - Indications for prescribing antibiotics (no positive dynamics or worsening of the patient's condition).
* The decrease in the total score (the sum of scores for each symptom) according to the LTM Scale (0-15), - Patients self-assessment (VAS; 0-10) scale of local manifestations of tonsillitis at the V 2, V 3 and V 4 in comparison with the 1-st visit. - Decrease in temperature in the armpit at the V 2 and V 3 compared to the Visit 1. - Self-evaluation of the patient's quality of life. - Duration of NSAID administration

Statistical endpoints:

The main criterion (main variable):

- the decrease in the severity of each symptom (complaint) that is part of the scale of tonsillitis manifestations, up to 1 point or less. This variable is dichotomous, with the categories "treatment effective" and "treatment not effective": Treatment is effective - reducing the severity of each symptom (complaint) that is part of the Local Tonsillitis Manifestation Scale (0-15),of tonsillitis manifestations, up to 1 point or less in the evaluation stages. Absence of indications for prescribing antibacterial therapy Treatment is not effective - the condition is given for the category "therapy is effective" is not met.

Secondary variables:

* The decrease in the severity of the symptoms of the underlying disease, at the V 2, V 3 and V 4 visits compared to the 1-st visit.
* The decrease in the total score (the sum of scores for each symptom) according to the scale of local manifestations of tonsillitis at the V 2, V 3 and V 4 in comparison with the 1-st visit.
* Decrease in temperature in the armpit at the 2-nd and 3-rd visits compared to the 1-st visit.
* Patient's self-assessment of the quality of life (every day).
* Duration of antipyretics administration. Statistical analysis is performed by a statistician and includes descriptions of patients (included, completed and withdrawn), adverse events and reactions, analysis of efficacy in each group, comparison of efficacy between groups, safety assessment, and tolerability in each group. It is planned to use the criteria of Shapiro-Wilk, Mann-Whitney (U).

Biometry: Patients with acute tonsillitis (N = 200): Age: 6-12 years old. The main group (n = 100). The control group (n = 100).

ELIGIBILITY:
Inclusion Criteria:

* Children (males/females), 6 - 12 years old, with severe acute tonsillitis.
* Possibility to initiate therapy within 72 hours since the onset of the disease symptoms.
* Score 4-5 according to McIsaac Scale.
* Patient's and (or) one of his/her parents' willingness and ability to fulfil the requirements of the Study Protocol.
* Signed informed consent of the patient and (or) his/her parents for participation in the study.

Exclusion Criteria:

* Score -1 to 3 according to McIsaac Scale.
* Indication for hospitalization, including:

  * purulent complications (peritonsillar abscess and others);
  * severe general condition.
* Indication for immediate initiation of systemic antibiotic therapy
* patients at risk of developing severe complications, including e.g. clinically relevant concomitant diseases of heart, lungs, kidneys, liver, neuromuscular apparatus, cancer diseases, immunosuppression, diabetes mellitus, cystic fibrosis.
* suspected infectious mononucleosis (by clinical signs);
* use of systemic antibacterial or antifungal agents, systemic glucocorticosteroids, cytostatics, immunomodulatory drugs, "interferons" or interferon derivatives during the last 14 days prior to inclusion;
* presence of haemorrhagic or pronounced necrotic process in oral cavity or pharynx, including the lymphoid ring.
* Intolerability or individual hypersensitivity to any of the study drug ingredients and the reference treatment scheme.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
- Changes in the severity of each symptom (complaint). | Day 1; 3; 5; 10; 28
  - Changes in the severity of each symptom (complaint; 0 - 4 points per symptom) that is part of the Acute tonsilitis severity scale of tonsillitis manifestations, up to 1 point or less. This variable is dichotomous, with the categories "treatment effective" and "treatment not effective".

CONTACTS AND LOCATIONS:
Overall Officials: Vasyl Popovych, Principal Investigator — Ivano-Frankivsk NMU
Locations (1):
- Ivano-Frankivsk National Medical University, Ivano-Frankivsk, Ivano-Frankivsk Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdulkerimov KT, Kartashova KI, Davydov RS, Abdulkerimov ZK, Kolesnikova AV, Yusupova DR. [The comparative evaluation of the effectiveness of the treatment of the patients presenting with the sub-compensated form of chronic tonsillitis making use of the antiseptic herbal medicinal product in the combination with the standard conservative therapy: the results of the open randomized study]. Vestn Otorinolaringol. 2018;83(3):45-49. doi: 10.17116/otorino201883345. Russian. PMID 29953055
- See also: Effectiveness and tolerability of Tonsilgon® N in the treatment of recurrent upper res-piratory tract infections in children: A non-interventional study in Russia, Clinical Phy-toscience (2016) — http://link.springer.com/article/10.1186/s40816-016-0020-9

DOCUMENTS (3):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04537819/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04537819/SAP_001.pdf
  • Informed Consent Form (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04537819/ICF_002.pdf